CLINICAL TRIAL: NCT00048217
Title: A Rollover Study to Provide Chronic T-1249 to Patients Who Completed Study T1249-102
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trimeris (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: T1249-105
Record Dates: First submitted 2002-10-28; First posted 2002-10-30 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — peptide T1249

INTERVENTIONS:
Drug: T-1249

SUMMARY:
Patients who complete study T1249-102 (must be currently failing a T-20 containing regimen to participate in this study) will receive T-1249 at a dose of 200mg daily in combination with a background antiretroviral regimen for 96 weeks. Only patients that participated in study T1249-102 can participate in study T1249-105.

ELIGIBILITY:
Inclusion Criteria:

* Completion T1249-102;
* Currently failing a T-20 containing regimen

Exclusion Criteria:

* Non-completion of T1249-102.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Trimeris, Durham, North Carolina, United States